CLINICAL TRIAL: NCT04544059
Title: Lenalidomide Plus R-CHOP for CNS Relapse Prophylaxis in Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Ru Feng, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NFDLBCL-CNS1
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: diffuse large b cell lymphoma; central nervous system; Lenalidomide
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide orally 25 mg per day was administered on days 1 through 10 of each cycle and delivered concomitantly with standard dose R-CHOP-21 regimen (rituximab 375 mg/m2, cyclophosphamide 750 mg/m2, doxorubicin 50 mg/m2 or Liposome doxorubicin 30mg/m2, vincristine 1.4 mg/m2 [capped at 2.0 mg], all on day 1; prednisone 100 mg per day on days 1 through 5). All patients received aspirin 100mg per day prophylaxis throughout, unless they were on therapeutic dose warfarin or low molecular weight heparin for intercurrent conditions. The treatment continued for a maximum of six to eight cycles or until disease progression. Tumor lysis prophylaxis, antiemetics, and supportive care were standard of care.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide orally 25 mg per day was administered on days 1 through 10 of each cycle and delivered concomitantly with standard dose R-CHOP-21 regimen (rituximab 375 mg/m2, cyclophosphamide 750 mg/m2, doxorubicin 50 mg/m2 or Liposome doxorubicin 30mg/m2, vincristine 1.4 mg/m2 [capped at 2.0 mg], all on day 1; prednisone 100 mg per day on days 1 through 5). All patients received aspirin 100mg per day prophylaxis throughout, unless they were on therapeutic dose warfarin or low molecular weight heparin for intercurrent conditions. The treatment continued for a maximum of six to eight cycles or until disease progression. Tumor lysis prophylaxis, antiemetics, and supportive care were standard of care.

SUMMARY:
This is an open-label, multicenter, phase 2 trial to explore the efficacy and safety of the combination of lenalidomide and R-CHOP for preventing the CNS relapse in the high-risk diffuse large B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

age 18-72 years histologically confirmed DLBCL High risk for CNS recurrence: CNS-IPI:4-6 or involvement of testicular, kidneys or adrenal glands.

No pregnancy plans during treatment

Exclusion Criteria:

Evidence of CNS involvement, Transformed lymphoma, Primary mediastinal B-cell lymphoma EBV+DLBCL, Secondary malignancy, HIV positive, Creatinine > 2.0 mg/dl Intending to hematopoietic stem cell transplantation history of severe thrombus Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The 2-year central nervous system relapse rates | two year
  The 2-year central nervous system relapse rates

SECONDARY OUTCOMES:
The 2-year overall survival | two year
  The 2-year overall survival
The 2-year progression-free survival | two year
  The 2-year progression-free survival
Incidence of treatment-emergent adverse events | two year
  Adverse events were classified as defined by the National Cancer Institute Common Toxicity Criteria, version 2. Safety evaluations were focused especially on neurological symptoms and the development of deep venous thrombosis (DVT).

CONTACTS AND LOCATIONS:
Overall Officials: Ru Feng, Principal Investigator — Department of Hematology, Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang hospital, Guangzhou, Guangdong, China